CLINICAL TRIAL: NCT05634122
Title: Efficacy of Acceptance and Commitment Therapy in Patients Scheduled for Lumbar Spine Surgery (SPINE-ACT Project)
Brief Title: Efficacy of ACT in Patients Scheduled for Lumbar Spine Surgery
Acronym: SPINE-ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Juan Ramon Castaño, Principal Investigator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/9998/I
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Randomized Controlled Trial
MeSH Terms: interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: parallel-group, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + Acceptance and Commitment Therapy (ACT) (Experimental): This therapy is based, as the name implies, on the acceptance (not avoidance) of negative experiences as a coping strategy, and on committing to life values or objectives. ACT has been used for various conditions, including chronic pain. Since avoidance is a strategy frequently used by patients suffering from pain, the application of this therapy seems very appropriate. In fact, it has been proven that patients who accept their pain more are those who score lower in pain intensity, have less negative emotions and enjoy a better quality of life.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Treatment as Usual (TAU) (Active Comparator): Standard care. The standard treatment would generally be pharmacological to address chronic pain, adjusted to the symptomatic profile of each patient.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Group treatment protocol of 8 weeks of 90 minutes sessions Session 1: Presentation of the general ACT therapy concept. Session 2: Value analysis I. Session 3: Value analysis II. Session 4: Value analysis third Session 5: Values and feelings. Session 6: Drink one direction. Session 7: Dare and change. Session 8: Ready to act with ACT. Treatment as usual (TAU) Standard pharmacological treatment for patients with chronic pain.
  Arms: TAU + Acceptance and Commitment Therapy (ACT)
Behavioral: Treatment as Usual (TAU) — Standard pharmacological treatment for patients with chronic pain
  Arms: Treatment as Usual (TAU)

SUMMARY:
Objectives: (1) To analyze the effectiveness of adding a group-based form of Acceptance and Commitment Therapy (ACT) to the treatment as usual (TAU) for preoperative patients diagnosed with degenerative lumbar pathology plus psychosocial risk factors related to post-surgical chronic pain at baseline and after psychological treatment. (2) To examine the effectiveness of ACT on the improvement of pain interference, pain-related and behavioral variables in degenerative lumbar pathology preoperative patients after lumbar spine surgery in comparison with TAU. (3) To measure the proximal and distal effects of ACT in preoperative patients with degenerative lumbar pathology who had the surgery after ACT program completion in comparison with proximal and distal TAU surgery effects on pain related variables.

Method: A 12-month randomized controlled trial (RCT) will be conducted at Hospital del Mar (Barcelona). Only those preoperative degenerative lumbar pathology patients with psychosocial risk factors for chronic post-surgical pain will be randomized to pre-surgical ACT group or to TAU. Evaluations will be completed before treatment (baseline), after ACT therapy (3 months), a first follow-up (6 months from baseline alias 3 months after surgery), second follow-up (9 months from baseline alias 6 months after surgery), and final follow-up (15 months from baseline alias 12 months from surgery).

Participants: 80 adult preoperative patients with degenerative lumbar pathology plus psychosocial risk factors related to post-surgical chronic pain will be randomly assigned to two arms: ACT + TAU vs TAU.

Primary outcome: Pain interference. Secondary outcomes: pain intensity, pain catastrophising, pain acceptance, pain disability, kinesiophobia, depression symptoms, anxiety symptoms, psychological flexibility, and quality of life.

Main statistical analyses: Intention-to-Treat analyses that will include all participants who undergo random allocation, using multiple imputation to replace missing values. General linear mixed-effects models will be performed using Restricted Maximum Likelihood to estimate the parameters. Calculation of between-groups effect sizes using Cohen's d and of the number-needed-to-treat.

DETAILED DESCRIPTION:
The Spine-ACT project's main objective is to determine the effectiveness of adding to the standard care (TAU) of preoperative patients with degenerative lumbar pathology plus psychosocial risk factors related to post-surgical chronic pain, a group-based form of ACT. In this regard, assessing patients' results after surgery at proximal or distal improvement on pain-related variables compared with TAU surgery patients would be addressed. The Spine-ACT project will assess the usefulness of ACT therapy applied before surgery to improve pain-related variables and quality of life in preoperative degenerative lumbar pathology patients with psychosocial risk factors of developing chronic or post-surgical pain. This project will significantly expand the limited knowledge available about preoperative pain-related improvement through ACT therapy and how this psychological therapy could prevent post-surgical chronic pain. Thus, it is expected that ACT therapy can improve the various pain-related and quality-of-life variables in developing chronic pain in preoperative patients diagnosed with degenerative lumbar pathology plus psychosocial risk factors of post-surgical chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 80 years
* Possess an adequate understanding of Spanish or Catalan
* Meet the diagnostic criteria for lumbar pain/degenerative lumbar pathology candidates for surgical treatment.

  * Diagnoses:

    1. Lumbar canal stenosis.
    2. Foraminal stenosis.
    3. Lumbar spondylolisthesis.
    4. Lumbar degenerative disc disease.
    5. Degenerative scoliosis.
    6. Lumbar kyphosis.
  * Procedures:

Laminectomy. Foraminoplasty. Laminectomy and posterior arthrodesis. previous arthrodesis.

* Presence of psychosocial risk factors for chronic post-surgical pain:

  * Mild-moderate anxiety/depression symptoms (HADS hospital anxiety and depression sub-scales≥11, see measurement instruments section) and/or
  * Presence of catastrophizing (PCS catastrophizing scale (0-52) ≥24, see measurement instruments section), and/or
  * Kinesiophobia base ≥27, see measurement instruments section)
* Have an internet connection on a mobile phone, tablet, computer, etc. to be able to carry out group psychological therapy online.
* Give authorization by signing an informed consent

Exclusion Criteria:

* Cognitive impairment that in the clinician's judgment prevents you from participating in therapy
* Presenting chronic pain not related to the diagnosis of low back pain that is a candidate for surgical treatment
* NOT present psychosocial risk factors for chronic post-surgical pain (see inclusion criteria: anxiety, catastrophizing, depression, kinesiophobia)
* Patients in litigation or who are pending legal claims for compensation
* Severe or decompensated psychiatric disorder (depression, schizophrenia, bipolar disorder, personality disorder) that in the clinician's judgment prevents you from participating in therapy
* Suicidal ideation
* Consumption of toxic substances in abuse/dependence, except for smoking
* Patients with a language barrier (Spanish/Catalan)
* Patients who do not authorize it voluntarily and do not want to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Through study completion, an average of 2 years
  It is a questionnaire that assesses chronic pain in a multidimensional way. It provides information on the intensity of the pain and on the degree of interference in the functioning and daily activities of the patients. It has 11 items. The first 4 items evaluate the intensity of pain in the last 24 hours. Subsequently, 7 items that report the degree of involvement of chronic pain in various areas of the person's functioning are evaluated. The higher the score in the areas of the questionnaire, the greater the intensity of perceived pain, as well as the greater degree of involvement of chronic pain in the functioning of the person in the various areas explored

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 2 years
  A scale of 14 items was created to assess symptoms of anxiety and depression. The total score ranges from 0 to 42, and each subscale (HADS-Anxiety and HADS-Depression) includes 7 items with scores ranging from 0 to 21. Higher scores indicate higher symptom severity.
Pain Catastrophising Scale (PCS) | Through study completion, an average of 2 years
  The scale of 13 items comprises three dimensions: rumination over pain, magnification of pain, and helplessness in the ace of pain symptoms. The PCS total score and subscale scores are computed as the sum of ratings for each item. This study used the total score, which can vary from 0 to 52 with higher scores indicating greater pain catastrophizing.
Psychological Inflexibility in Pain Scale (PIPS) | Through study completion, an average of 2 years
  12-item scale that assesses psychological inflexibility in patients with pain and includes two factors: avoidance and cognitive fusion with pain. For this study, only the total score is used; it ranges from 12 to 84, with higher scores indicating higher level of psychological inflexibility.
Tampa Kinesiophobia Scale (TSK-11SV) | Through study completion, an average of 2 years
  It is a questionnaire that allows us to measure the fear of moving or being injured/(re)injured, in patients with pain. The final score can be at least 11 and a maximum of 44 points; the higher the score, the higher the degree of kinesiophobia. It is considered that a score ≥18 is already indicative of a fear of movement, which increases in severity as the score increases.
Chronic Pain Acceptance Questionnaire (CPAQ-20) | Through study completion, an average of 2 years
  It consists of 20 items organized in a factorial structure of two subscales. The maximum possible total score is 120, so that higher scores indicate a higher level of the acceptance construct in the process.
Short Form 12 Health Survey (SF-12) | Through study completion, an average of 2 years
  This scale includes measures of health-related quality of life. It is made up of a subset of 12 items, with 8 dimensions, and 2 summative components (physical and mental). The items are coded, added, and transformed into a scale that ranges from 0 (the worst state of health for that dimension) to 100 (the best state of health).
Oswestry Low Back Pain Disability Scale (OLBPDQ) | Through study completion, an average of 2 years
  The scale consists of 10 questions with 6 response possibilities each. The total score, expressed as a percentage (0 to 100%), is obtained as the sum of the estimates for each element divided by the maximum possible score multiplied by 100. High values describe greater functional limitations.

OTHER OUTCOMES:
Socio-demographic questionnaire | Baseline
  Gender, date of birth, marital status, living arrangements, educational level and employ-ment status.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Montes-Pérez, PhD, Study Director — Parc Salut Mar; Víctor Pérez-Solà, PhD, Study Director — Parc Salut Mar; Luis Miguel Martín-López, PhD, Study Chair — Parc Salut Mar; Alejandro Del Arco-Churruca, PhD, Study Director — Parc Salut Mar; Jesús Lafuente Baraza, PhD, Study Chair — Parc Salut Mar; Juan V. Luciano, PhD, Study Director — Parc Sanitari Sant Joan de Déu; Juan Ramón Castaño-Asins, MD, Principal Investigator — Parc Salut Mar
Locations (1):
- Parc Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No